CLINICAL TRIAL: NCT05386355
Title: Improving Pediatric COVID-19 Vaccine Uptake Using an mHealth Tool: a Randomized, Controlled Trial
Brief Title: Improving Pediatric COVID-19 Vaccine Uptake Using an mHealth Tool
Acronym: MoVeUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IDeA States Pediatric Clinical Trials Network (Network)
Collaborators: National Institutes of Health (NIH) (NIH); University of Nebraska (Other); University of Montana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 273761; U24OD024957 (NIH)
Record Dates: First submitted 2022-05-19; First posted 2022-05-23 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: COVID-19 Vaccines; Telemedicine; Vaccine Hesitancy; Pediatric ALL
Keywords: COVID-19; COVID-19 vaccination; Pediatric COVID-19 vaccination; mobile health; mHealth
MeSH Terms: conditions — Vaccination Hesitancy; Precursor Cell Lymphoblastic Leukemia-Lymphoma; COVID-19

STUDY DESIGN:
Intervention Model Description: The study will use a 1:1 parallel design at the caregiver level to assign caregivers to the intervention (Vaccine Uptake app) or the control (General Health app) arm. The study team will stratify randomization by participating clinic and in varying block of participants using a permuted design. Randomization will occur after enrollment and before the baseline assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine Uptake App (Experimental): 24-week (8 weeks with weekly push notifications; 2 monthly push notifications for 2 months [1 notification per month]; 8 weeks without) exposure to a mobile phone application (app) designed to improve parental knowledge, attitudes, and self-efficacy regarding pediatric COVID-19 vaccination. The app will address logistical and motivational barriers to pediatric COVID-19 vaccination. Participants will also receive eight weekly nudges and 1 monthly nudge for 2 months (cues to action) regarding vaccinating their child that will be sent to participants via push notifications to their mobile devices. Through branching logic, users will access content tailored to their COVID-19 vaccine knowledge and confidence gaps, locality, degree of rural-urban primary residence, primary language (English/Spanish), race/ethnicity, and child's age.
  Interventions: Behavioral: COVID-19 Vaccine Uptake App
- General Health App (Active Comparator): 24-week (8 with weekly push notifications; 2 monthly push notifications for 2 months [1 notification per month]; 8 weeks without) exposure to a mobile phone app designed to provide information on general pediatric health and infection prevention and mitigation strategies based on recommendations from the American Academy of Pediatrics (AAP) and the Centers for Disease Control and Prevention (CDC). Eight weekly nudges and 1 monthly nudge for 2 months regarding these topics will be sent to participants via push notifications to their mobile devices.
  Interventions: Other: General Health App

INTERVENTIONS:
Behavioral: COVID-19 Vaccine Uptake App — A mHealth mobile application (app) that will provide educational and logistical information about the COVID-19 vaccination for children. The target audience will be parents of unvaccinated children.
  Arms: Vaccine Uptake App
Other: General Health App — A mobile application (app) that will provide general pediatric health and infection prevention and mitigation strategies.
  Arms: General Health App

SUMMARY:
This study will determine the effectiveness of a vaccine communication mobile health app on parental decisions to vaccinate their children against coronavirus disease 2019 (COVID-19).

The hypothesis is that unvaccinated children of caregivers assigned to the Vaccine Uptake app will be more likely to achieve COVID-19 vaccine series completion than those children whose caregivers are assigned to the General Health app.

DETAILED DESCRIPTION:
This is a site-level block-randomized trial. The study population is Custodial parents/caregivers with ≥1 child eligible for COVID-19 vaccination who has not yet received the vaccine at the time of study enrollment.

The primary objective is to determine the effect of a parent-facing, vaccination decision-making mobile health (mHealth) tool on children's COVID-19 vaccine series completion. The endpoint of this objective is the proportion of children who complete COVID-19 vaccination, as verified in state, clinic, or participant-held records.

Secondary Objective 1 is to determine the effect of a parent-facing, vaccination decision-making mHealth tool on children's COVID-19 vaccine series initiation. The endpoint of this objective is the proportion of children who receive ≥1 dose of the COVID-19 vaccination series, as verified in state, clinic, or participant-held records

Secondary Objective 2 is to determine the effect of a parent-facing, vaccination decision-making mHealth tool on parental attitude toward pediatric COVID-19 vaccination. The endpoint of this objective is the change in enrolled parent/caregiver domain scores from baseline to week 16 on the modified World Health Organization (WHO) Strategic Advisory Group of Experts on Immunization (SAGE) Vaccine Hesitancy Scale adapted for the COVID-19 Vaccine.

Enrolling sites will recruit participants. These sites will collaborate with outpatient practices within Environmental influences on Child Health Outcomes (ECHO) Institutional Development Award (IDeA) States Pediatric Clinical Trials Network (ISPCTN) states that provide primary care services to children (<18 years old). Sites will serve a population base of at least 40% Medicaid/uninsured children, <60% non-Hispanic White children, or >40% of families residing in rural communities. Sites are encouraged, but not required, to have a high Spanish-speaking population.

Study interventions are a Vaccine Uptake App and General Health App. The Vaccine Uptake App will include 24-week (8 weeks with weekly push notifications; 2 monthly push notifications for 2 months [1 notification per month]; 8 weeks without) exposure to a mobile phone application (app) designed to improve parental knowledge, attitudes, and self-efficacy regarding pediatric COVID-19 vaccination. The app will address logistical and motivational barriers to pediatric COVID-19 vaccination. Participants will also receive eight weekly nudges and 1 monthly nudge for 2 months (cues to action) regarding vaccinating their child that will be sent to participants via push notifications to their mobile devices. Through branching logic, users will access content tailored to their COVID-19 vaccine knowledge and confidence gaps, locality, degree of rural-urban primary residence, primary language (English/Spanish), race/ethnicity, and child's age.

The General Health App will include 24-week (8 weeks with weekly push notifications; 2 monthly push notifications for 2 months [1 notification per month]; 8 weeks without) exposure to a mobile phone app designed to provide information on general pediatric health and infection prevention and mitigation strategies based on recommendations from the American Academy of Pediatrics (AAP) and the Centers for Disease Control and Prevention (CDC). Nudges regarding these topics will be sent to participants via push notifications to their mobile devices.

The study duration is 24 months (6 months study start-up; up to 8 months rolling enrollment; 7 months final participants' completion; 3 months analysis). Participant duration is 27 weeks.

ELIGIBILITY:
Parent/Caregiver Inclusion Criteria:

* Age of majority, as defined by the state of residency
* Access to a mobile device that can store and run the study app for 24 weeks. Devices that can run the app include mobile phones and tablets running Android or iOS operating systems
* Able to speak and read in English or Spanish
* Be a parent/caregiver with primary medical decision-making and legal authority to consent to vaccination decisions for at least one child who meets the child inclusion criteria

Child Inclusion Criteria:

* Age 6 months to less than age of majority, as defined by the child's state of residence
* Has not received any doses of COVID-19 vaccine based on parent/caregiver report
* Eligible to receive COVID-19 vaccine
* Patient at a participating clinic

Parent/Caregiver Exclusion Criteria:

* Has only a child or children with known contraindication to all COVID-19 vaccines
* Has only a child or children whose other parent/caregiver is already a current or past participant in the study
* Has a child or children enrolled in any other COVID-19 vaccine study of any kind
* Past or present participation in a COVID-19 vaccine or behavioral trial
* Has a cognitive impairment that limits their ability to engage with the app content and/or make medical decisions regarding vaccination, based on the site investigator's assessment and local human subjects research policies

Child Exclusion Criteria:

* Not a patient of a participating clinic
* Prior receipt of least one dose of COVID-19 vaccine
* Receiving or scheduled to receive COVID-19 vaccination at the time of parental consent
* Known medical contraindication to all COVID-19 vaccines
* Ineligible to receive COVID-19 vaccine
* Prior or current participation in a COVID-19 vaccine study of any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1934 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell J. McCulloh, MD, Principal Investigator — University of Nebraska; Ellen Kerns, PhD, Principal Investigator — University of Nebraska; Paul Darden, MD, Principal Investigator — University of Arkansas; Songthip T Ounpraseuth, PhD, Study Director — University of Arkansas
Locations (15):
- United States (15):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - Nemours Children's Health, Wilmington, Delaware
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Children's Research Institute, Louisville, Kentucky
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Clinic, Lebanon, New Hampshire
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
We will conduct this trial in accordance with the following publication and data sharing policies and regulations:
  * NIH Public Access Policy. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication.
  * ECHO ISPCTN Publications and Presentations Policy. It ensures accurate, responsible, and efficient communication of findings from ECHO ISPCTN clinical trials.
  * NIH Data Sharing Policy and the policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Resulting Information Submission Rule. Other researchers may request data from this trial by contacting Jeannette Lee, Ph.D., at the ISPCTN Data Coordinating and Operations Center (DCOC).
Supporting Information: SAP, ICF
Time Frame: Per data sharing polices of NIH and the ISPCTN
Access Criteria: to be announced

REFERENCES:
- [Derived] McCulloh RJ, Darden PM, Snowden J, Ounpraseuth S, Lee J, Clarke M, Newcomer SR, Fu L, Hubberd D, Baldner J, Garza M, Kerns E. Improving pediatric COVID-19 vaccine uptake using an mHealth tool (MoVeUp): study protocol for a randomized, controlled trial. Trials. 2022 Oct 28;23(1):911. doi: 10.1186/s13063-022-06819-3. PMID 36307830
- [Derived] McCulloh RJ, Darden P, Snowden J, Ounpraseuth S, Lee J, Clarke M, Newcomer SR, Fu L, Hubberd D, Baldner J, Garza M, Kerns E. Improving pediatric COVID-19 vaccine uptake using an mHealth tool (MoVeUP): a randomized, controlled trial. Res Sq [Preprint]. 2022 Oct 10:rs.3.rs-2070396. doi: 10.21203/rs.3.rs-2070396/v1. PMID 36238712

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol enrollment number of 727 represent the total number of parents/caregivers that were enrolled and randomized. For the study the unit of randomization is the parent/caregiver. The primary and secondary outcomes of interest, vaccine series completion and vaccine series initiation, were collected at the children level. Among these 727 parents/caregivers, there was a total of 1,207 children enrolled.
Groups:
- Vaccine Uptake App: Parents/Caregivers; Vaccine Uptake App: Children: 24-week (8 weeks with weekly push notifications; 2 monthly push notifications for 2 months [1 notification per month]; 8 weeks without) exposure to a mobile phone application (app) designed to improve parental knowledge, attitudes, and self-efficacy regarding pediatric COVID-19 vaccination. The app will address logistical and motivational barriers to pediatric COVID-19 vaccination. Participants will also receive eight weekly nudges and 1 monthly nudge for 2 months (cues to action) regarding vaccinating their child that will be sent to participants via push notifications to their mobile devices. Through branching logic, users will access content tailored to their COVID-19 vaccine knowledge and confidence gaps, locality, degree of rural-urban primary residence, primary language (English/Spanish), race/ethnicity, and child's age.
  COVID-19 Vaccine Uptake App: A mHealth mobile application (app) that will provide educational and logistical information about the COVID-19 vaccination for children. The target audience will be parents of unvaccinated children.
- General Health App: Parents/Caregivers; General Health App: Children: 24-week (8 with weekly push notifications; 2 monthly push notifications for 2 months [1 notification per month]; 8 weeks without) exposure to a mobile phone app designed to provide information on general pediatric health and infection prevention and mitigation strategies based on recommendations from the American Academy of Pediatrics (AAP) and the Centers for Disease Control and Prevention (CDC). Eight weekly nudges and 1 monthly nudge for 2 months regarding these topics will be sent to participants via push notifications to their mobile devices.
  General Health App: A mobile application (app) that will provide general pediatric health and infection prevention and mitigation strategies.
Period: Overall Study
Arm/Group | Vaccine Uptake App: Parents/Caregivers | General Health App: Parents/Caregivers | Vaccine Uptake App: Children | General Health App: Children
Started | 361 (This represents the number of parent/caregiver that were randomized to the Vaccine Uptake App cohort. This included 612 children.) | 366 (This represents the number of parent/caregiver that were randomized to the General Health App cohort. This included 595 children.) | 612 (This represents the number of children among the parents/caregivers that were randomized to the Vaccine Uptake App cohort.) | 595 (This represents the number of children among the parents/caregivers that were randomized to the General Health App cohort.)
Completed | 360 | 365 | 611 | 594
Not Completed | 1 | 1 | 1 | 1
Not completed — Each group had an ineligible child (i.e., one over 18 years old and one less than 6-months old). | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: A total of 727 parent/caregiver were enrolled and randomized. Two participants were ineligible (1 from Vaccine Uptake App and 1 from General Health App) since one had a child over 18 years old and the other had a child < 6 months old. Therefore, the final analytical sample size was 725 parent/caregiver (Vaccine Uptake App N = 360 and General Health App N = 365) and 1205 children (Vaccine Uptake App N = 611 and General Health App N = 594).
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine Uptake App: Parents/Caregivers | General Health App: Parents/Caregivers | Vaccine Uptake App: Children | General Health App: Children | Total
Number analyzed (Participants) | 360 | 365 | 611 | 594 | 1930
Age, Customized [Count of Participants; unit: Participants] — Measure Description: Age was not collected for parent/caregiver. Population: Measure Description: Age was not collected for parent/caregiver.
  Participants
    Age, Customized: number analyzed (Participants) | 0 | 0 | 611 | 594 | 1205
    Age, Customized: 6 months - 5 years |  |  | 273 | 271 | 544
    Age, Customized: 5 - 11 years |  |  | 243 | 224 | 467
    Age, Customized: 12 - 17 years |  |  | 95 | 99 | 194
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The number analyzed in the row represents the number of parent/caregiver and children in each of the four defined groups (Vaccine Uptake App Parents/Caregivers; General Health Parent/Caregivers; Vaccine Uptake Children; General Health Children). However, the total overall number represents the sum of parent/caregiver plus children for each row.
  Participants
    Male | 18 | 25 | 326 | 300 | 669
    Female | 341 | 340 | 285 | 294 | 1260
    Not listed/prefer not to answer | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed in the row represents the number of parent/caregiver and children in each of the four defined groups (Vaccine Uptake App Parents/Caregivers; General Health Parent/Caregivers; Vaccine Uptake Children; General Health Children). However, the total overall number represents the sum of parent/caregiver plus children for each row.
  Participants
    Hispanic or Latino | 61 | 64 | 115 | 95 | 335
    Not Hispanic or Latino | 298 | 300 | 495 | 499 | 1592
    Unknown or Not Reported | 1 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed in the row represents the number of parent/caregiver and children in each of the four defined groups (Vaccine Uptake App Parents/Caregivers; General Health Parent/Caregivers; Vaccine Uptake Children; General Health Children). However, the total overall number represents the sum of parent/caregiver plus children for each row.
  Participants
    American Indian or Alaska Native | 2 | 10 | 5 | 9 | 26
    Asian | 0 | 4 | 0 | 6 | 10
    Native Hawaiian or Other Pacific Islander | 2 | 0 | 3 | 1 | 6
    Black or African American | 130 | 132 | 222 | 222 | 706
    White | 179 | 167 | 282 | 258 | 886
    More than one race | 17 | 19 | 52 | 50 | 138
    Unknown or Not Reported | 30 | 33 | 47 | 48 | 158
Caregiver Education [Count of Participants; unit: Participants] — Population: For the education measure, only 512 parent/caregivers completed the baseline survey (General Health App N = 255 and Vaccine Uptake App N = 257).
  Participants
    <= High school or GED completed: number analyzed (Participants) | 257 | 255 | 0 | 0 | 512
    <= High school or GED completed | 94 | 60 | 0 | 0 | 154
    Some college/technical/vocational: number analyzed (Participants) | 257 | 255 | 0 | 0 | 512
    Some college/technical/vocational | 85 | 117 | 0 | 0 | 202
    Bachelor's degree: number analyzed (Participants) | 257 | 255 | 0 | 0 | 512
    Bachelor's degree | 45 | 45 | 0 | 0 | 90
    Master's/Doctoral: number analyzed (Participants) | 257 | 255 | 0 | 0 | 512
    Master's/Doctoral | 23 | 23 | 0 | 0 | 46
    Unknown/prefer not to answer: number analyzed (Participants) | 257 | 255 | 0 | 0 | 512
    Unknown/prefer not to answer | 5 | 6 | 0 | 0 | 11
    Missing: number analyzed (Participants) | 257 | 255 | 0 | 0 | 512
    Missing | 5 | 4 | 0 | 0 | 9
Number of Children [Median (Inter-Quartile Range); unit: Number of Children] — Population: The number analyzed in the row represents the number of parent/caregiver since this measure is only relevant at the parent/caregiver level.
  Number of Children
    number analyzed (Participants) | 360 | 365 | 0 | 0 | 725
    (all) | 1 [1 to 2] | 1 [1 to 2] |  |  | 1 [1 to 2]
Rurality (self-reported) [Count of Participants; unit: Participants] — Population: The number analyzed in the row represents the number of parent/caregiver since rurality is only reported at the parent/caregiver level.
  Participants
    Yes: number analyzed (Participants) | 360 | 365 | 0 | 0 | 725
    Yes | 115 | 134 |  |  | 249
    No: number analyzed (Participants) | 360 | 365 | 0 | 0 | 725
    No | 245 | 231 |  |  | 476

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Children Who Complete COVID-19 Vaccination, as Verified in State, Clinic, or Participant-held Records
Description: Initiation and completion of the COVID-19 vaccine series during the 24-week intervention period. Vaccine series completion will be per ACIP guidance for the vaccine product. For children who receive a product that requires more than 2 doses for the primary series, receipt of up to 3 doses will be considered complete. Vaccine doses will be valid if given within 24-week study intervention. Additional doses for primary series completion will be valid if they are in accordance with ACIP-recommended interval minus a 4-day grace period. There will be no maximum interval between valid doses. An incorrect second vaccine product (i.e., mixed series) will be invalid. The statistical team will use a mixed model with the binomial distribution and the logit link to compare the two intervention groups and the proportions of children who complete COVID-19 vaccination, using a site random effect and controlling for clustering by caregiver.
Time Frame: Week 24
Population: Randomization was at the parent/caregiver level; however, the unit of analysis for the primary (vaccine series completion) and secondary (vaccine series initiation) are at the children level. There were total of 1205 children (Vaccine Uptake N=611 and General Health N=595). Among the 1205, the vaccine completion outcome contained 11 missing observations (5 from Vaccine Uptake and 6 from General Health group).
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Uptake App: Children | General Health App: Children
Number analyzed (Participants) | 606 | 588
Participants | 13 | 7
Statistical Analysis 1: Comparison: Vaccine Uptake App: Children vs General Health App: Children; A mixed-effect Poisson regression with robust variance estimation was used report the adjusted RR with 95% CI accounting for the clinic-specific random intercepts. Given the small number of COVID-19 vaccination completion, we were unable to account for children nested with parent/caregiver or adjusting for covariates; Test type: Superiority; Risk Ratio (RR) = 1.79, 95% CI 2-sided [0.59 to 5.35] — The General Health App is the reference group

2. Secondary Outcome: Proportion of Children Who Receive ≥1 Dose of the COVID-19 Vaccination Series, as Verified in State, Clinic, or Participant-held Records
Description: For each vaccine-eligible child, this secondary endpoint will be defined as whether or not the child initiates the COVID-19 vaccine series during the 16 weeks of study participation. Vaccine series initiation will be receipt of at least 1 valid dose of any COVID-19 vaccine product. Vaccine doses for series initiation will only be valid for study purposes if given within the 16 weeks of study participation. The statistical team will use a mixed model with the binomial distribution and the logit link to compare the two intervention groups with respect to the proportions of children who initiate COVID-19 vaccination, using site as a random effect and controlling for clustering by caregiver.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Uptake App: Children | General Health App: Children
Number analyzed (Participants) | 606 | 588
Participants | 22 | 25
Statistical Analysis 1: Comparison: Vaccine Uptake App: Children vs General Health App: Children; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.42 to 1.65] — The General Health App is the reference group

3. Secondary Outcome: Change in Enrolled Parent/Caregiver Domain Scores From Baseline to Immediately Post-intervention on the Modified WHO SAGE Vaccine Hesitancy Scale Adapted for the COVID-19 Vaccine
Description: The Strategic Advisory Group of Experts on Immunization (SAGE) working group on vaccine hesitancy developed a vaccine hesitancy measure, the Vaccine Hesitancy Scale (VHS). The study team will evaluate parental attitude toward pediatric COVID-19 vaccination by using the vaccine hesitancy questionnaire that includes ten statements with ordinal responses using a 5-point Likert scale (1=strongly disagree,...,5=strongly agree).
  A composite vaccine hesitancy score was computed based on the sum of the 10 items after reverse coding items 1, 2, 3, 4, 6, 7, and 8 (range of 10 to 50). The reverse coding allowed for directionality uniformed across the 10 items; therefore, higher composite score indicated more hesitancy overall. We report summary statistics including means and standard deviation at baseline and week 16. A linear mixed mode was used to account for parent/caregivers nested within clinics and allow adjustment for baseline SAGE composite score.
Time Frame: 16 weeks
Population: The vaccine hesitancy secondary outcome is analyzed at the parent/caregiver level. Among the 725 parent/caregiver randomized, a total of 512 parent/caregiver completed the baseline survey.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Vaccine Uptake App: Parents/Caregivers | General Health App: Parents/Caregivers
Number analyzed (Participants) | 257 | 255
score on a scale | 23.33 [22.25 to 24.16] | 23.10 [22.27 to 23.93]
Statistical Analysis 1: Comparison: Vaccine Uptake App: Parents/Caregivers vs General Health App: Parents/Caregivers; Test type: Superiority; p = 0.638, Mixed Models Analysis; The analytical method was based on a linear mixed model adjusting for baseline SAGE vaccine hesitancy composite scores and random clinic effect; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-1.19 to 0.73]

ADVERSE EVENTS:
Time Frame: 32 weeks
Description: The unit of randomization was at the parent/caregiver level. We randomized 727 parent/caregiver (2 participants were ineligible with one participant having an only child over 18 years old while another participant had an only child under 6 months old). The unit of analysis is at the children level. There were a total of 1205 children (General Health App N=594 and Vaccine Uptake N=611). There were no adverse events reported at the parent/caregiver level.
Arm/Group | General Health App: Children | Vaccine Uptake App: Children | General Health App: Parents/Caregivers | Vaccine Uptake App: Parents/Caregivers
All-Cause Mortality (participants affected / at risk) | 0/594 | 0/611 | 0/365 | 0/360
Serious Adverse Events (participants affected / at risk) | 0/594 | 0/611 | 0/365 | 0/360
Other Adverse Events (participants affected / at risk) | 1/594 | 0/611 | 0/365 | 0/360
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General Health App: Children (N=594) | Vaccine Uptake App: Children (N=611) | General Health App: Parents/Caregivers (N=365) | Vaccine Uptake App: Parents/Caregivers (N=360)
Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — New onset diabetes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT05386355/Prot_001.pdf
  • Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT05386355/SAP_002.pdf
  • Informed Consent Form (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT05386355/ICF_000.pdf